CLINICAL TRIAL: NCT03502993
Title: Personalised Risk Assessment in Febrile Illness to Optimise Real-life Management Across the European Union (PERFORM)
Acronym: PERFORM
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Liverpool (Other); University of Newcastle Upon-Tyne (Other); Erasmus Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); National and Kapodistrian University of Athens (Other); Stichting Katholieke Universiteit (Other); University of Graz (Other); University of Ljubljana (Other); Riga Stradins University (Other); Medical Research Council Unit, The Gambia (Other); Ludwig-Maximilians - University of Munich (Other); University of Bern (Other); University of Oxford (Other); University Hospital, Paris (Other); University of Santiago de Compostela (Other); Servicio Gallego de Salud (Other Government); BioMérieux (Industry); Micropathology Ltd, University of Warwick (Industry)
Responsible Party: Sponsor
Other Study IDs: REC ref: 16/LO/1684; BIVA studies (Other: Imperial College London)
Record Dates: First submitted 2018-03-27; First posted 2018-04-19 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Fever; Infection; Inflammation
Keywords: children
MeSH Terms: conditions — Fever; Infections; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, nasopharyngeal aspirate/throat swab, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BIVA studies - children with fever and/or suspected infection: A minimum of 3,000 children will be recruited to the BIVA-ED (Biomarker Validation in Emergency Department) study, in order to capture sufficient children with confirmed bacterial infection. Additional children with less common febrile illnesses will also be recruited: 500 critically ill (BIVA-PIC); 200 at high-risk of bacterial illness through primary or secondary immunodeficiency (BIVA-HR); 150 with an inflammatory diagnosis, whose initial presentation is difficult to discriminate from bacterial infection (BIVA-INF). Samples collected from recruits in the BIVA studies will be used for the validation of biomarkers (clinical, proteomic and transcriptomic biomarkers) for diagnosis of febrile illness, including markers of bacterial and viral infection (confirmed by culture and/or molecular microbiology) and inflammatory conditions.
  Interventions: Diagnostic Test: Validation of biomarker
- BIVA studies - control children without fever or suspicion of infection: Afebrile children <18 years (16 years depending in the setting) of age who are having blood tests for reasons other than for investigation of infectious or inflammatory illness or whom parents give consent for bloods taken for research purposes. Controls may have a range of clinical presentations including co-morbidities without infection. One set of samples will be taken from controls, no follow up data or samples taken.
  Interventions: Diagnostic Test: Validation of biomarker

INTERVENTIONS:
Diagnostic Test: Validation of biomarker

SUMMARY:
Childhood fever is a prevalent problem. Most febrile children who visit hospital improve without treatment, but a minority require treatment, and a few will have severe disease. The investigators want to improve the diagnosis and management of febrile children by developing tests to distinguish between bacterial and viral disease so that antibiotic treatment can be initiated promptly and only when required. Judicious and prudent use of antibiotics will reduce the likelihood of developing resistant organisms and save treatment costs.

The investigators will prospectively recruit acutely febrile children presenting to hospital, collecting research samples for validation of biomarkers, in combination with clinical phenotypic markers and host genetic markers (BIVA-studies).

Any febrile child newborn to under 18 presenting to hospital will be eligible for recruitment. The study will last 5 years.

DETAILED DESCRIPTION:
The problem to be addressed:

Fever is among the commonest symptoms for which parents consult health care providers worldwide. Distinction between life-threatening bacterial infection and viral infection is clinically difficult, and many children worldwide receive unnecessary antibiotic treatment, or undergo invasive investigations and hospitalization, whilst bacterial infection is missed in others.

Objective:

The investigators aim to validate biomarkers that will identify children with bacterial infection, viral infection and inflammatory syndromes, using whole-blood RNA expression, proteomic and metabolomics signatures. The investigators aim to assess how efficacious these biomarkers would be if they formed the basis of a diagnostic test.

Design:

The investigators will use established case-control groups of febrile children presenting to hospital, recruited across Europe as part of previous (and current) ethically-approved studies, to discover signatures of febrile illness. The investigators will validate these signatures in samples prospectively collected from children as part of this observational study.

The investigators will use prospective, observational BIVA studies to recruit febrile children with infectious and inflammatory diseases in order to validate diagnostic biomarkers. The investigators will also recruit non-febrile controls in order to discover and validate disease-specific biomarkers and to understand their biological significance.

STUDY SIZE at least 4000 febrile children;

PROCEDURES;

Informed consent using age appropriate patient/parent/guardian information sheets will be taken from parents (or from children aged 16 and over), assent will be taken from the child under the age of 16 (if appropriate).

Routine clinical and laboratory data and research samples from three timepoints (presentation, 48 hours after presentation, 28 days after admission). If patients present to hospital with fever on subsequent occasions, clinical data will be recorded and further research samples will be taken at those times.

Samples; Blood, urine, stool (in the case of gastroenteritis), nasopharyngeal/throat swab

CONTROLS:

The investigators will collect samples from age-matched control patients will not have had a febrile illness, major trauma or vaccination within the previous three weeks and who are having routine blood sampling for reasons other than investigation of infectious or inflammatory disease.

Control children may include critically ill children without infection or those with healthcare associated infections.

ELIGIBILITY:
Inclusion Criteria:

* All children <18 years with fever >38ºC, or a history of fever (within 3 days), in whom the attending clinician determines the need for blood sampling or whom parents give consent for bloods taken for research purposes
* All children <18 years suspected of infection, including the full spectrum of disease severity and co-morbidities.
* Afebrile control children who are having blood tests for reasons other than for investigation of infectious or inflammatory illness.

Exclusion Criteria:

* Children from whom parent/legal guardian signed consent is not received
* For healthy control children only: febrile illness or vaccination within the last 3 weeks.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with fever >38ºC, or a history of fever (within 3 days) who requires a blood test for clinical reasons or consents for research bloods to be taken,
Sampling Method: Probability Sample
Enrollment: 7247 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levin, Study Chair — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Habgood-Coote D, Wilson C, Shimizu C, Barendregt AM, Philipsen R, Galassini R, Calle IR, Workman L, Agyeman PKA, Ferwerda G, Anderson ST, van den Berg JM, Emonts M, Carrol ED, Fink CG, de Groot R, Hibberd ML, Kanegaye J, Nicol MP, Paulus S, Pollard AJ, Salas A, Secka F, Schlapbach LJ, Tremoulet AH, Walther M, Zenz W; Pediatric Emergency Medicine Kawasaki Disease Research Group (PEMKDRG); UK Kawasaki Genetics consortium; GENDRES consortium; EUCLIDS consortium; PERFORM consortium; Van der Flier M, Zar HJ, Kuijpers T, Burns JC, Martinon-Torres F, Wright VJ, Coin LJM, Cunnington AJ, Herberg JA, Levin M, Kaforou M. Diagnosis of childhood febrile illness using a multi-class blood RNA molecular signature. Med. 2023 Sep 8;4(9):635-654.e5. doi: 10.1016/j.medj.2023.06.007. Epub 2023 Aug 18. PMID 37597512
- [Derived] Hartman SJF, Upadhyay PJ, Hagedoorn NN, Mathot RAA, Moll HA, van der Flier M, Schreuder MF, Bruggemann RJ, Knibbe CA, de Wildt SN. Current Ceftriaxone Dose Recommendations are Adequate for Most Critically Ill Children: Results of a Population Pharmacokinetic Modeling and Simulation Study. Clin Pharmacokinet. 2021 Oct;60(10):1361-1372. doi: 10.1007/s40262-021-01035-9. Epub 2021 May 26. PMID 34036552
- See also: publications and conference proceedings pertaining to PERFORM - BIVA studies — https://cordis.europa.eu/project/id/668303/results

RESULTS

PARTICIPANT FLOW:
Groups:
- BIVA Studies: A minimum of 3,000 children will be recruited to the BIVA-ED study, in order to capture sufficient children with confirmed bacterial infection. Additional children with less common febrile illnesses will also be recruited: 500 critically ill (BIVA-PIC); 200 at high-risk of bacterial illness through primary or secondary immunodeficiency (BIVA-HR); 150 with an inflammatory diagnosis, whose initial presentation is difficult to discriminate from bacterial infection (BIVA-INF). Samples collected from recruits in the BIVA studies will be used for the validation of biomarkers (clinical, proteomic and transcriptomic biomarkers) for diagnosis of febrile illness, including markers of bacterial and viral infection (confirmed by culture and/or molecular microbiology) and inflammatory conditions.
  Validation of biomarker
- Control Children Without Fever or Suspicion of Infection: Children attending hospital for reasons other than for investigation of febrile illness or suspicion of infection
Period: Overall Study
Arm/Group | BIVA Studies | Control Children Without Fever or Suspicion of Infection
Started | 5957 | 1290
Completed | 5957 | 1290
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Controls for BIVA Studies: Age-matched control patients will not have had a febrile illness, major trauma or vaccination within the previous three weeks and who are having routine blood sampling for reasons other than investigation of infectious or inflammatory disease.
  Control children may include critically ill children without infection or those with healthcare associated infections.
  Where data was incomplete, patients were not included in the analysis - therefore the number analysed is not always 1290
- Total: Total of all reporting groups
Arm/Group | BIVA Studies | Controls for BIVA Studies | Total
Number analyzed (Participants) | 5957 | 1290 | 7247
Age, Customized [Median (Inter-Quartile Range); unit: years] — Population: Participants excluded from age analysis if data missing or incomplete
  years
    age on presentation: number analyzed (Participants) | 5924 | 1231 | 7155
    age on presentation | 4.57 [1.68 to 9.74] | 9.64 [5.02 to 13.42] | 5.32 [1.93 to 10.82]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants excluded from sex analysis if data missing or incomplete
  Participants
    number analyzed (Participants) | 5957 | 1239 | 7196
    Female | 2638 | 544 | 3182
    Male | 3319 | 695 | 4014
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants excluded from race/ethnicity analysis if data missing or incomplete
  Participants
    reported ethnicity/race: number analyzed (Participants) | 5870 | 1237 | 7107
    reported ethnicity/race: North/Mid/East European | 2999 | 718 | 3717
    reported ethnicity/race: South European | 1209 | 384 | 1593
    reported ethnicity/race: Mandinka | 194 | 0 | 194
    reported ethnicity/race: unknown | 146 | 0 | 146
    reported ethnicity/race: Roma European | 115 | 2 | 117
    reported ethnicity/race: Mixed | 110 | 17 | 127
    reported ethnicity/race: FULA | 97 | 0 | 97
    reported ethnicity/race: Gambian | 93 | 0 | 93
    reported ethnicity/race: Arabian Peninsula/Arab Middle East | 91 | 9 | 100
    reported ethnicity/race: West Asian | 88 | 11 | 99
    reported ethnicity/race: WOLOF | 70 | 0 | 70
    reported ethnicity/race: North African | 67 | 7 | 74
    reported ethnicity/race: East Asian | 61 | 21 | 82
    reported ethnicity/race: other | 46 | 9 | 55
    reported ethnicity/race: Serahule | 45 | 0 | 45
    reported ethnicity/race: Afro-Carribean | 31 | 5 | 36
    reported ethnicity/race: South East Asian | 30 | 1 | 31
    reported ethnicity/race: Native South American | 18 | 3 | 21
    reported ethnicity/race: Other African | 13 | 10 | 23
    reported ethnicity/race: Other EU | 8 | 1 | 9
    reported ethnicity/race: Other Asian | 3 | 3 | 6
    reported ethnicity/race: South Asian Nepal | 3 | 0 | 3
    reported ethnicity/race: Jewish | 7 | 0 | 7
    reported ethnicity/race: South Asian Indian, Pakistani, Bangladeshi | 170 | 20 | 190
    reported ethnicity/race: Subsaharan Africa | 112 | 9 | 121
    reported ethnicity/race: Turkish | 44 | 7 | 51
Co-morbidities leading to increased infection risk, BIVA studies [Number; unit: participants] — Population: Participants excluded from Co-morbidities leading to increased infection risk, BIVA studies analysis if data missing or incomplete
  participants
    number analyzed (Participants) | 5957 | 1250 | 7207
    (all) | 446 | 43 | 489

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically-assigned Retrospective Phenotype
Description: Clinically-assigned retrospective phenotype, according to the cause of illness
Time Frame: Participants were monitored for outcome throughout their stay in hospital, and received follow-up review at 10 days
Population: Number of children with definite bacterial illness assessed by positive blood culture and/or positive culture of sample from sterile site
Measure: Count of Participants; unit: Participants
Arm/Group | BIVA Studies | Controls for BIVA Studies
Number analyzed (Participants) | 5952 | 1290
Participants | 655 | 0

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse outcomes throughout their stay in hospital and monitored upto follow up period of 10 days
Description: Observational study; outcome (death)
Groups:
- Healthy Controls: Children attending hospital for reasons other than investigation of febrile illness or suspicion of infection
Arm/Group | BIVA Studies | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 50/5957 | 0/1290
Serious Adverse Events (participants affected / at risk) | 120/5957 | 0/1290
Other Adverse Events (participants affected / at risk) | 0/5957 | 0/1290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIVA Studies (N=5957) | Healthy Controls (N=1290)
Sepsis syndrome (Blood and lymphatic system disorders) | 120 (120) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03502993/Prot_SAP_000.pdf
  • Informed Consent Form (2016-06-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT03502993/ICF_001.pdf